CLINICAL TRIAL: NCT04826055
Title: tp Make the Length of the Biliary Limb as a Percentage From the Small Intestine Rather Than Fixed Length in Loop Bypass Surgery for Morbid Obesity
Brief Title: Biliary Limb as a Percentage From the Small Intestine Rather Than Fixed Length in Loop Bypass Surgery for Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor and consultant of general surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fac.med 21.17
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Morbid
Keywords: biliary limb length in bypass bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- loop bypass with fixed biliary limb length (Active Comparator): in all loop bypass procedures we will don't count the total length of small intestine and make the biliary limb as a fixed from total small intestine length as mentioned in literature
  Interventions: Other: biliary limb as fixed length
- loop bypass with a biliary limb is a percentage of the small intestine (Experimental): in all loop bypass procedures we count the total length of small intestine and make the biliary limb as a percentage from total small intestine length rather than fixed length
  Interventions: Other: biliary limb as a percentage from small intestine length

INTERVENTIONS:
Other: biliary limb as fixed length — n all loop bypass procedures we will don't count the total length of small intestine and make the biliary limb as a fixed from total small intestine length as mentioned in literature
  Arms: loop bypass with fixed biliary limb length
Other: biliary limb as a percentage from small intestine length — in all loop bypass procedures we count the total length of small intestine and make the biliary limb as a percentage from total small intestine length rather than fixed length
  Arms: loop bypass with a biliary limb is a percentage of the small intestine

SUMMARY:
in all loop bypass bariatric procedure (mini gastric bypass & single anastomosis sleeve jejunal bypass), biliary limb is fixed length. we do it as a percentage from total small intestine length rather than fixed length

DETAILED DESCRIPTION:
in all loop bypass bariatric procedure (mini gastric bypass & single anastomosis sleeve jejunal bypass), biliary limb is fixed length we count the length of small intestine and do it as a percentage from total small intestine length rather than fixed length

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 or more than 35 with comorbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 50
* patients with BMI less than 35
* patient with previous upper abdominal surgery either for obesity or other diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
effect on weight loss | one year
  the effect on weight loss
effect on nutritional deficiency | 1 year
  the effect on nutritional deficiency

SECONDARY OUTCOMES:
operative time | 6 hours
  operative time from skin incision to skin closure
effect on obesity comorbidities | 1 year
  the effect on improvement of obesity related comorbidities
early complications | 30 days
  the operative and postoperative 30 days complications
late complications | 1 year
  the late reported complications

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Minya, Egypt